CLINICAL TRIAL: NCT04712500
Title: A Single-Center, Randomized, Open-Label, Two-Sequence, Two-Period Crossover Study in Healthy Non-Elderly Chinese Subjects to Evaluate the Food Effect on the Pharmacokinetics of AND017 Following Oral Single-Dose Administration
Brief Title: A Food-Effect Study of AND017 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AND017-CN-101
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AND017: Fasted - Fed (Experimental): Subjects were randomized to receive single dose of AND017 under fasted condition in Period 1 and under fed condition in Period 2
  Interventions: Drug: AND017
- AND017: Fed - Fasted (Experimental): Subjects were randomized to receive single dose of AND017 under fed condition in Period 1 and under fasted condition in Period 2
  Interventions: Drug: AND017

INTERVENTIONS:
Drug: AND017 — AND017 oral capsule

SUMMARY:
The purpose of this phase I study is to evaluate the food effect on the PKs of AND017 following oral single-dose administration in healthy non-elderly Chinese subjects.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, two-sequence, two-period crossover study in healthy non-elderly Chinese subjects to evaluate the food effect on the pharmacokinetics, as well as PD and safety of AND017 following oral single-dose administration

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 19.0~26.0 kg/m2 (both inclusive); Body weight ≥50 kg for male, and ≥45 kg for female.
2. Healthy participants having no clinical significant abnormalities of examinations during screening period and at the time of informed consent
3. Have no pregnancy plan in the next six months and are willing to take effective contraceptive methods.

Exclusion Criteria:

1. Allergic constitution or has a history of allergy to AND017 capsule and its excipient;
2. Subjects with low blood pressure or a risk of low blood pressure: systolic pressure <90 mmHg, diastolic pressure<60 mmHg.
3. Subjects with difficulty in venous blood sampling;
4. Subjects with a history of drug abuse within the past five years or who have abused drug within the past three months before screening;
5. Subjects smoking more than five cigarettes a day or nicotine dependent within the past three months before screening;
6. Subjects drinking alcohol more than 14 U/week within the past six months or used any alcohol products in two days pre-dose;
7. Subjects that have received any medication within the past 4 weeks pre-dose;
8. Subjects that have taken food or drink that has the potential to induce or inhibit drug metabolizing enzymes in the liver within one-week pre-dose;
9. Subjects that have taken any food or drink that contains or can be metabolized to caffeine or xanthine from 48 hours pre-dose to the last PK or PD blood sampling;
10. Subjects with diseases or factors of clinical abnormalities that need to be excluded, including but not limited to the nervous system, cardiovascular system, kidney, liver, gastrointestinal, respiratory system, metabolism, and skeletal system diseases, or other factors that may affect drug absorption, distribution, metabolism and excretion;
11. Subjects that have used HIF-PHIs within the past one year;
12. Subjects positive in HIV-Ab, HBsAg or HBeAg, or HCV-Ab, TP-Ab;
13. Subjects that have participated in any other clinical trials within the past three months pre-dose in the study;
14. Female subjects of childbearing age who are pregnant, lactating, or planning pregnancy; or have a positive in pregnancy test during the study;
15. Subjects with a history of blood donation or had a blood loss more than 400 mL within three months before screening;
16. Subjects that have special requirements on diet and cannot follow the dietary program indicated in the study;
17. Subjects that are unable to comply with research requirements or with any factors are considered not suitable for participating in the study according to the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 6, 0-72 hours post-dose
  Maximum Observed Plasma Concentration for AND017
AUC0-inf | Day 1 and Day 6, 0-72 hours post-dose
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time for AND017

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD PhD, Study Director — Kind Pharmaceuticals LLC
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No